CLINICAL TRIAL: NCT05937178
Title: A Real-world Study of Optimizing Nucleotide-analogues-based Treatment for Chronic Hepatitis B
Brief Title: Real-world Study Optimizing Nucleotide-analogues
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other); Anhui Provincial Hospital (Other Government); Beijing YouAn Hospital (Other); Peking University People's Hospital (Other); Peking University First Hospital (Other); Xiamen Hospital of Traditional Chinese Medicine (Other); First Affiliated Hospital of Fujian Medical University (Other); LanZhou University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); First Affiliated Hospital of Guangxi Medical University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Hainan General Hospital (Other); Hebei Medical University Third Hospital (Other); The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); Henan Provincial People's Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Tongji Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Renmin Hospital of Wuhan University (Other); Central South University (Other); Xiangya Hospital of Central South University (Other); The First Hospital of Jilin University (Other); the Second Hospital of Nangjing (Unknown); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The First Affiliated Hospital with Nanjing Medical University (Other); The Affiliated Hospital of Xuzhou Medical University (Other); The First Affiliated Hospital of Nanchang University (Other); Shengjing Hospital (Other); Qingdao Sixth People's Hospital (Unknown); Shandong Provincial Hospital (Other Government); The Second Hospital of Shandong University (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Tang-Du Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Ruijin Hospital (Other); West China Hospital (Other); Tianjin Second People's Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); The First People's Hospital of Yunnan (Other); Shulan (Hangzhou) Hospital (Other); Zhejiang University (Other); Southwest Hospital, China (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Other Study IDs: REASON
Record Dates: First submitted 2023-06-28; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Recommend to initiate treatment in 2022 Chinese Guideline, but not in 2019 Chinese Guideline: Untreated population who does not be recommended to initiate treatment in 2022 Chinese Guideline, but not in 2019 Chinese Guideline. The initate treatment is to receive a first-line nucleos(t)ide analogue, i.e., entecavir, tenofovir disoproxil, or tenofovir alafenamide, tenofovir amibufenamide
  Interventions: Drug: ETV/TAF/TDF/TMF
- Recommend to initiate treatment in 2019 and 2022 Chinese Guideline, but not in AASLD/EASL guidelines: Untreated population will receive a first-line nucleos(t)ide analogue , i.e., entecavir, tenofovir disoproxil, or tenofovir alafenamide, tenofovir amibufenamide, and the population should meet the conditions that are recommended to initiate treatment in 2019 and 2022 Chinese guideline, but not in AASLD/EASL guidelines
  Interventions: Drug: ETV/TAF/TDF/TMF
- Treatment experienced and with partial response: Treatment experienced population who has received a first-line nucleos(t)ide analogue(NA) as monotherapy at least 48 weeks, i.e., entecavir, tenofovir disoproxil, or tenofovir alafenamide, tenofovir amibufenamide, and has partial response to NA. They will continue the original therpay or plans to change the therapy (e.g. switch another first-line NA, add-on another first-line NA, switch another first-line NA and add-on peginterferon alpha)
  Interventions: Drug: ETV/TAF/TDF/TMF/IFN

INTERVENTIONS:
Drug: ETV/TAF/TDF/TMF/IFN — peginterferon alpha or nucleos(t)ide alone are decided by patients' doctors according to their conditions, instead of extra interventions brought by the study
  Groups: Treatment experienced and with partial response
Drug: ETV/TAF/TDF/TMF — peginterferon alpha or nucleos(t)ide alone are decided by patients' doctors according to their conditions, instead of extra interventions brought by the study
  Groups: Recommend to initiate treatment in 2019 and 2022 Chinese Guideline, but not in AASLD/EASL guidelines; Recommend to initiate treatment in 2022 Chinese Guideline, but not in 2019 Chinese Guideline

SUMMARY:
The goal of this multicenter, observational, prospective study is to observe and compare different anti-viral treatment strategies in a real-world cohort of patients with CHB managed in routine clinical settings in China. The main questions it aims to answer are:

1. To evaluate the benefits of initiating first-line nucleos(t)ide analogue in patients with chronic HBV infection who are recommended in the updated Chinese Guideline 2022, but not recommended in the Chinese Guideline 2019.
2. To evaluate the Chinese Guideline recommends initiation of treatment, but at least one foreign authoritative guideline (eg. AASLD, EASL) does not recommend the benefit of initiating first-line nucleos(t)ide analogue in patients with chronic HBV infection who initiate treatment.
3. To compare the treatment effect of different alternatives with patients who have partial response after treatment with first-line nucleos(t)ide analogues.

DETAILED DESCRIPTION:
REASON is a multicenter, observational, prospective study to explore an optimal anti-viral treatment in a real-world cohort of patients with CHB managed in routine clinical settings in China. The study will enroll treatment-naïve or treatment-experienced patients ≥18 and ≤80 years of age with hepatitis B s antigen positive. The treatment-experienced patients must be treated with monotherapy ETV/TDF/TAF/TMF continuously for a minimum of 48 weeks before enrollment. The treatment of participants will be decided before the screening by doctors based on the situation and patient's intention. When eligible patients are included in this study, no extra intervention will be conducted and only clinical data are collected and observed. Participants will enter different observation groups when they meet the eligibility criteria of each group listed below: Group A：treatment-naive, and meeting the conditions that are recommended to initiate treatment in 2022 Chinese Guideline but not in 2019 Chinese Guideline; Group B：treatment-naive, meeting the conditions that are recommended to initiate treatment in both 2019 and 2022 Chinese guideline, but not in AASLD/EASL guidelines; Group C: treatment-experienced and with partial response. The primary efficacy endpoint was the proportion of patients with HBV DNA less than 20 IU/ml at 48 weeks, 96 weeks, and 144 weeks. Participants in all groups will be stratified by whether they initiate treatment in Group A and B, and by the treatment regimens in Group C. The primary safety outcome is the change from baseline in the Estimated Glomerular Filtration Rate by the Cockcroft-Gault Formula (eGFR-CG) at 48 weeks, 96 weeks, and 144 weeks. The secondary outcomes including HBsAg loss, HBsAg seroconversion, HBeAg loss, HBeAg seroconversion, fibrosis regression and progression, and liver-related events, which will be measured at each follow-up visit. The follow-up time course of this study will be 3 years.

ELIGIBILITY:
Inclusion Criteria:

* CHB defined as positive hepatitis B surface antigen at least 6 months, or HBV-related histological changes within 1 year if HBsAg positive less than 6 months.
* Age between 18-80 years.
* Patient who reads and signs informed consent.
* Meet any conditions of the group listed below

Group A-naïve and meeting the conditions that are recommended to initiate treatment in 2022 Chinese Guideline, but not in 2019 Chinese Guideline (observe-plan to treat or control-plan to follow-up) :

A. HBV DNA positive, ALT is continuously upper limit of normal (male 30 U/L, female 19 U/L) B. HBeAg positive, HBV DNA≤2×10^7 IU/ml; HBeAg negative, HBV DNA≥2×10^3 IU/ml C. Meet any of the conditions listed below

1. Age>30 years, and have a family history of cirrhosis or HCC, TE indicates no significant fibrosis;
2. Family history of cirrhosis or HCC, and ≤30 years, TE indicates no significant fibrosis;
3. TE indicates significant fibrosis, and ≤30 years, without family history of cirrhosis or HCC

Group B-naïve and meeting the conditions that are recommended to initiate treatment in both 2019 and 2022 Chinese Guidelines, but not in EASL or AASLD guideline (observe-plan to treat or control-plan to follow-up) :

A. Without cirrhosis, HBV DNA≤2000 IU/ml, ALT>1 ULN； B. Without cirrhosis, HBV DNA>2000 IU/ml, 1 ULN<ALT≤2 ULN； C. Without cirrhosis, normal ALT, >30 years, have a family history of cirrhosis or HCC, or TE indicates significant fibrosis; D. Without cirrhosis, HBV DNA 20-2000 IU/ml Group C-experienced and partial response (1. switch another first-line NA; 2. add-on another first-line NA; 3. switch another first-line NA and add-on peginterferon alpha; 4. continue the original plan) Treatment experienced patient who has received a first-line nucleos(t)ide analogue(NA) monotherapy for at least 48 weeks, i.e., entecavir, tenofovir disoproxil or tenofovir alafenamide, tenofovir amibufenamide, and has partial response. They plan to continue or change the therapy

Exclusion Criteria:

* Have poor compliance;
* Received contraindicated concomitant drugs (subjects receiving prohibited drugs will need at least 30 days of washing out period) and known hypersensitivity reactions to the study drug, metabolites, or formulated excipients;
* Any other clinical symptoms or previous treatment that the investigator considers that the individual subject is not suitable for this study or cannot comply with the administration requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis B will receive the first-line antiviral therapy
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with HBV DNA <20 IU/ml | Week 48
  The primary efficacy endpoint was the proportion of patients with HBV DNA <20 IU/ml at each follow-up time point, as determined by high-sensitivity PCR
The proportion of patients with HBV DNA <20 IU/ml | Week 96
  The primary efficacy endpoint was the proportion of patients with HBV DNA <20 IU/ml at each follow-up time point, as determined by high-sensitivity PCR
The proportion of patients with HBV DNA <20 IU/ml | Week 144
  The primary efficacy endpoint was the proportion of patients with HBV DNA <20 IU/ml at each follow-up time point, as determined by high-sensitivity PCR
Change from baseline in Estimated Glomerular Filtration Rate by the Cockcroft-Gault Formula (eGFR-CG) | Baseline
  Change from baseline in Estimated Glomerular Filtration Rate by the Cockcroft-Gault Formula (eGFR-CG) at each follow-up time point
Change from baseline in Estimated Glomerular Filtration Rate by the Cockcroft-Gault Formula (eGFR-CG) | Week 48
  Change from baseline in Estimated Glomerular Filtration Rate by the Cockcroft-Gault Formula (eGFR-CG) at each follow-up time point
Change from baseline in Estimated Glomerular Filtration Rate by the Cockcroft-Gault Formula (eGFR-CG) | Week 96
  Change from baseline in Estimated Glomerular Filtration Rate by the Cockcroft-Gault Formula (eGFR-CG) at each follow-up time point
Change from baseline in Estimated Glomerular Filtration Rate by the Cockcroft-Gault Formula (eGFR-CG) | Week 144
  Change from baseline in Estimated Glomerular Filtration Rate by the Cockcroft-Gault Formula (eGFR-CG) at each follow-up time point

SECONDARY OUTCOMES:
Proportion of participants with Normal Alanine Aminotransferase (ALT) | Week 48, Week 96 and Week 144
  Proportion of participants with Normal Alanine Aminotransferase (ALT) at each follow-up time point
Proportion of participants with Hepatitis B s Antigen (HBsAg) Loss | Week 48, Week 96 and Week 144
  Proportion of participants with Hepatitis B s Antigen (HBsAg) Loss at each follow-up time point
Proportion of participants with Hepatitis B s Antigen (HBeAg) Loss | Week 48, Week 96 and Week 144
  Proportion of participants with Hepatitis B s Antigen (HBeAg) Loss at each follow-up time point
Proportion of participants with seroconversion to Hepatitis B s Antigen (HBsAg) | Week 48, Week 96 and Week 144
  Proportion of participants with seroconversion to Hepatitis B s Antigen (HBsAg) at each follow-up time point
Proportion of participants with seroconversion to Hepatitis B e Antigen (HBeAg) | Week 48, Week 96 and Week 144
  Proportion of participants with seroconversion to Hepatitis B e Antigen (HBeAg) at each follow-up time point
Proportion of participants with fibrosis regression and progression | Week 48, Week 96 and Week 144
  Proportion of participants with fibrosis regression and progression at each follow-up time point
Rate of liver-related events | Week 48, Week 96 and Week 144
  Rate of liver-related events (HCC, decompensation cirrhosis, death) at each follow-up time point

CONTACTS AND LOCATIONS:
Overall Officials: Wenghong Zhang, MD, Principal Investigator — Huashan Hospital; Jiming Zhang, MD, Principal Investigator — Huashan Hospital; Feng S, MD, Study Chair — Huashan Hospital; Qiran Zhang, MD, Study Director — Huashan Hospital
Locations (44):
- China (44):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing YouAn Hospita, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - the Southwest Hospital of AMU, Chongqing, Chongqing Municipality
  - First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Xiamen Hospital of Traditional Chinese Medicine, Xiamen, Fujian
  - the First Hospital of Lanzhou University, Lanzhou, Gansu
  - First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Affiliated Hospital Of Guizhou Medical University, Guiyang, Guizhou
  - The Second Affiliated Hospital of Harbin Medical University, Ha’erbin, Ha'erbin
  - Hainan General Hospital, Haikou, Hainan
  - the Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Tongji Hospital, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - the Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - the Second Hospital of Nangjing, Nanjing, Jiangsu
  - the Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - the First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - the First Bethune Hospital Of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Tangdu Hospital, The Fourth Military Medical University, Xi'an, Shaanxi
  - the First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - The Second Hospital of Shandong University, Jinan, Shandong
  - No. 6 People's Hospital of Qingdao, Qingdao, Shandong
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Second People's Hospital, Tianjin, Tianjin Municipality
  - Third Affiliated Hospital, Sun Yat-Sen University, Meizhou, Xiamen
  - Xinjiang Uygur Autonomous Region Hospital of Traditional Chinese Medicine, Ürümqi, Xinjiang Uygur Autonomous Region
  - First People's Hospital of Yunnan Province, Kunming, Yunnan
  - Shulan (Hangzhou) Hospital, Hangzhou, Zhejiang
  - Huashan Hospital, Shanghai

REFERENCES:
- [Background] Polaris Observatory Collaborators. Global prevalence, treatment, and prevention of hepatitis B virus infection in 2016: a modelling study. Lancet Gastroenterol Hepatol. 2018 Jun;3(6):383-403. doi: 10.1016/S2468-1253(18)30056-6. Epub 2018 Mar 27. PMID 29599078
- [Background] Chinese Society of Infectious Diseases, Chinese Medical Association; Chinese Society of Hepatology, Chinese Medical Association. [The guidelines of prevention and treatment for chronic hepatitis B (2019 version)]. Zhonghua Gan Zang Bing Za Zhi. 2019 Dec 20;27(12):938-961. doi: 10.3760/cma.j.issn.1007-3418.2019.12.007. Chinese. PMID 31941257
- [Background] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Background] Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on prevention, diagnosis, and treatment of chronic hepatitis B: AASLD 2018 hepatitis B guidance. Hepatology. 2018 Apr;67(4):1560-1599. doi: 10.1002/hep.29800. No abstract available. PMID 29405329
- [Background] Nassal M. HBV cccDNA: viral persistence reservoir and key obstacle for a cure of chronic hepatitis B. Gut. 2015 Dec;64(12):1972-84. doi: 10.1136/gutjnl-2015-309809. Epub 2015 Jun 5. PMID 26048673
- [Background] Agarwal K, Brunetto M, Seto WK, Lim YS, Fung S, Marcellin P, Ahn SH, Izumi N, Chuang WL, Bae H, Sharma M, Janssen HLA, Pan CQ, Celen MK, Furusyo N, Shalimar D, Yoon KT, Trinh H, Flaherty JF, Gaggar A, Lau AH, Cathcart AL, Lin L, Bhardwaj N, Suri V, Mani Subramanian G, Gane EJ, Buti M, Chan HLY; GS-US-320-0110; GS-US-320-0108 Investigators. 96 weeks treatment of tenofovir alafenamide vs. tenofovir disoproxil fumarate for hepatitis B virus infection. J Hepatol. 2018 Apr;68(4):672-681. doi: 10.1016/j.jhep.2017.11.039. Epub 2018 Jan 17. PMID 29756595
- [Background] Chinese Society of Infectious Disease Chinese Society of Hepatology; Chinese Medical Association. [The expert consensus on clinical cure (functional cure) of chronic hepatitis B]. Zhonghua Gan Zang Bing Za Zhi. 2019 Aug 20;27(8):594-603. doi: 10.3760/cma.j.issn.1007-3418.2019.08.003. Chinese. PMID 31594076
- [Background] Zhang L, Fan ZF, Liu DW, Zhou MG, Wang ZQ, Li M. [Trend analysis on the disease burden related to cirrhosis and other chronic liver diseases caused by hepatitis B, in China, from 1990 to 2016]. Zhonghua Liu Xing Bing Xue Za Zhi. 2020 Feb 10;41(2):173-177. doi: 10.3760/cma.j.issn.0254-6450.2020.02.007. Chinese. PMID 32164125
- [Background] Kim GA, Lim YS, An J, Lee D, Shim JH, Kim KM, Lee HC, Chung YH, Lee YS, Suh DJ. HBsAg seroclearance after nucleoside analogue therapy in patients with chronic hepatitis B: clinical outcomes and durability. Gut. 2014 Aug;63(8):1325-32. doi: 10.1136/gutjnl-2013-305517. Epub 2013 Oct 25. PMID 24162593
- [Background] Lim TH, Gane E, Moyes C, Borman B, Cunningham C. HBsAg loss in a New Zealand community study with 28-year follow-up: rates, predictors and long-term outcomes. Hepatol Int. 2016 Sep;10(5):829-37. doi: 10.1007/s12072-016-9709-6. Epub 2016 Mar 8. PMID 26957439
- [Background] Sinn DH, Kim SE, Kim BK, Kim JH, Choi MS. The risk of hepatocellular carcinoma among chronic hepatitis B virus-infected patients outside current treatment criteria. J Viral Hepat. 2019 Dec;26(12):1465-1472. doi: 10.1111/jvh.13185. Epub 2019 Aug 13. PMID 31332935
- [Background] ZHUANG H. Should chronic hepatitis B in the indeterminate phase be treated?[J]. J Clin Hepatol, 2021, 37(9): 2033-2036.
- [Background] Chinese Society of Hepatology, Chinese Medical Association. [Expert opinion on expanding anti-HBV treatment for chronic hepatitis B]. Zhonghua Gan Zang Bing Za Zhi. 2022 Feb 20;30(2):131-136. doi: 10.3760/cma.j.cn501113-20220209-00060. Chinese. PMID 35359064
- [Background] National Health and Family Planning Commission of the People's Republic of China. China Statistical Yearbook. Beijing: Peking Union Medical College Press, 2020.
- [Background] Wang G, Duan Z. Guidelines for Prevention and Treatment of Chronic Hepatitis B. J Clin Transl Hepatol. 2021 Oct 28;9(5):769-791. doi: 10.14218/JCTH.2021.00209. Epub 2021 Sep 28. PMID 34722192